CLINICAL TRIAL: NCT01547247
Title: Cap-assisted Water Immersion Versus Water Immersion Minimal Sedation Colonoscopy - a Prospective, Randomized, Single-center Trial
Brief Title: Cap-assisted Water Immersion Versus Water Immersion Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt MD, Principal Investigator, Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDC VN 03
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Colonoscopy
Keywords: colonoscopy; cap-assisted colonoscopy; water immersion colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cap-assisted water immersion colonoscopy (Experimental): Cap-fitted colonoscopy using purely water immersion during colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Interventions: Device: soft straight distal cap D-201-14304 Olympus attached to the tip of the colonoscope
- water immersion colonoscopy (Active Comparator): Standard colonoscopy without attached cap using purely water immersion during colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Interventions: Procedure: water immersion colonoscopy

INTERVENTIONS:
Device: soft straight distal cap D-201-14304 Olympus attached to the tip of the colonoscope — Colonoscopy with transparent cap attached to the tip of the colonoscope and water immersion during insertion phase and romm air insufflation during colonoscope withdrawal.
  Arms: cap-assisted water immersion colonoscopy
Procedure: water immersion colonoscopy — Colonoscopy without transparent cap using water immersion during insertion phase and romm air insufflation during colonoscope withdrawal.
  Arms: water immersion colonoscopy

SUMMARY:
Water immersion insertion has been documented to decrease procedure-related discomfort during colonoscopy. Cap attached to the colonoscope tip may improve insertion and shorten cecal intubation time. The investigators would like to assess whether combination of cap-fitted colonoscopy and water immersion insertion is feasible and safe method of diagnostic colonoscopy. The primary endpoint is cecal intubation time and the investigators suppose that the use of cap is able to shorten it significantly. Patient comfort during colonoscope insertion, water consumption, length of the scope while reaching the cecum, need for external compression, need for positioning of the patient and endoscopist´s difficulty with colonoscopy are assessed.

ELIGIBILITY:
Inclusion Criteria:

* outpatient diagnostic colonoscopy
* bowel prep with macrogolum
* initial 2 mg of midazolam i.v.
* signed informed consent form

Exclusion Criteria:

* planned therapeutic intervention
* colorectal surgery in history
* known inflammatory bowel disease or colorectal cancer
* refusal of sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Falt, MD, Principal Investigator — Digestive Diseases Center, Vitkovice Hospital
Locations (1):
- Digestive Diseases Center, Vitkovice Hospital, Ostrava, Czechia

REFERENCES:
- [Result] Falt P, Smajstrla V, Fojtik P, Liberda M, Kliment M, Tvrdik J, Urban O. Cap-assisted water immersion for minimal sedation colonoscopy: prospective, randomized, single-center trial. Dig Endosc. 2013 Jul;25(4):434-9. doi: 10.1111/j.1443-1661.2012.01402.x. Epub 2012 Dec 5. PMID 23808948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * recruitment period - between March and May 2012
  * consecutive patients referred to our endoscopic unit for diagnostic colonoscopy
Pre-assignment Details: * a total of 275 subjects assessed for eligibility
  * a total of 208 patients eandomized after exclusion of 67 due to not fulfilled inclusion criteria
  * a total of 196 subjects analyzed after exclusion of 12 patients (poor bowel preparation, IBD, malignant obstruction, protocol deviation, ischemic colitis)
Period: Overall Study
Arm/Group | Cap-assisted Water Immersion Colonoscopy | Water Immersion Colonoscopy
Started | 104 | 104
Completed | 98 | 98
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cap-assisted Water Immersion Colonoscopy | Water Immersion Colonoscopy | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 51 | 100
  >=65 years | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.0) | 58.2 (13.9) | 58.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 59 | 59 | 118
Region of Enrollment [Number; unit: participants]
  Czech Republic | 104 | 104 | 208

OUTCOME MEASURES:

1. Primary Outcome: Cecal Intubation Time
Description: The primary endpoint (cecal intubation time) was defined as a time between introduction of the colonoscope into the anus and reaching the cecum.
Time Frame: 3 months
Population: Statistical power was calculated for the primary endpoint. A sample size of 93 subjects per arm was calculated using two-tailed alfa 0.05, beta 0.2, assuming that difference 20 % in intubation times would have been clinically relevant.
Measure: Number (95% Confidence Interval); unit: minutes
Arm/Group | Cap-assisted Water Immersion Colonoscopy | Water Immersion Colonoscopy
Number analyzed (Participants) | 98 | 98
minutes | 6.9 [4.0 to 9.8] | 7.4 [3.2 to 11.6]

2. Secondary Outcome: Patient Comfort During Insertion Phase of the Colonoscopy
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Success Rate of Minimal Sedation Colonoscopy
Description: A successful minimal sedation colonoscopy was defined as reaching the cecum without switching to another insertion method and without additional sedation beyond the initial 2 mg of midazolam.
Time Frame: 3 months
Measure: Number; unit: percentage of all subjects in arm
Arm/Group | Cap-assisted Water Immersion Colonoscopy | Water Immersion Colonoscopy
Number analyzed (Participants) | 98 | 98
percentage of all subjects in arm | 91 | 91

ADVERSE EVENTS:
Arm/Group | Cap-assisted Water Immersion Colonoscopy | Water Immersion Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There were no complications recorded in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No